CLINICAL TRIAL: NCT05542381
Title: The Role of Loteprednol in Reducing Post-Intravitreal Injection Related Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Collaborators: Vistar Eye Center (Other)
Responsible Party: Principal Investigator, Vishak John, Retina Surgeon, Virginia Polytechnic Institute and State University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 22-514
Record Dates: First submitted 2022-09-01; First posted 2022-09-15 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-01

CONDITIONS: Age-Related Macular Degeneration
Keywords: Loteprednol; Loteprednol Etabonate Ophthalmic Suspension; Immunosuppressive Agents; Glucocorticoids; Immunologic Factors; Molecular Mechanisms of Pharmacological Action; Eye Diseases; Retinal Diseases; Anti-Inflammatory Agents; vascular endothelial growth factor; Intravitreal Injection; Post-Intravitreal Injection Pain
MeSH Terms: conditions — Macular Degeneration; Eye Diseases; Retinal Diseases | interventions — Loteprednol Etabonate; Lubricant Eye Drops

STUDY DESIGN:
Intervention Model Description: Double-blinded placebo-controlled design
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The study design is a double-blinded placebo-controlled experiment, as the patient and the investigator recording the pain scores will not know which treatment arm the patient is assigned to (negative control or experimental group).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Loteprednol (Experimental): 1 drop of Loteprednol is administered immediately after the intravitreal injection in this treatment arm.
  Interventions: Drug: Loteprednol Etabonate Ophthalmic Gel [Lotemax]
- Artificial tears (Placebo Comparator): 1 drop of artificial tears is administered immediately after the intravitreal injection in this treatment arm. This arm acts as a negative control.
  Interventions: Other: Refresh Lubricant Eye Drops [Artificial Tears]

INTERVENTIONS:
Drug: Loteprednol Etabonate Ophthalmic Gel [Lotemax] — Loteprednol (ophthalmic corticosteroid) will be stored in the clinic according to the instructions on the package. The vial will be stored upright between 15°-25°C (59°-77°F). In the clinic, the vial will be opened by the retina surgeon according to sterile procedure and administered (1 drop) by the surgeon immediately after the intravitreal injection.
  Arms: Loteprednol
Other: Refresh Lubricant Eye Drops [Artificial Tears] — REFRESH® Brand Lubricant Eye Drops are artificial tears. In the clinic, the vial will be opened by the retina surgeon according to sterile procedure and administered (1 drop) by the surgeon immediately after the intravitreal injection.
  Other Names: Refresh
  Arms: Artificial tears

SUMMARY:
Patients are already receiving an intravitreal injection as a standard of care, but they are consenting to receiving a loteprednol drop following the intravitreal injection. This clinical trial is studying the role of loteprednol (corticosteroid) in reducing pain following intravitreal injections for patients with age-related macular degeneration. As of now, there is no definitive pain management technique following intravitreal injections. Loteprednol is a corticosteroid widely used in ophthalmology to treat pain and inflammation, however, it has not been studied as a treatment for pain following intravitreal injections. Our overall goal is to manage pain to improve quality of care after intravitreal injections. Participants will be given either loteprednol, or artificial tears following one visit for an intravitreal injection to test how effective loteprednol is in pain reduction. Pain levels will be assessed by asking participants over the phone about their pain from a scale of 0 to 10 at three different times over a 1-week period. Artificial tear and medication usage will also be tracked over a 1-week period.

DETAILED DESCRIPTION:
Patients are already receiving an intravitreal injection as a standard of care for age-related macular degeneration, but they are consenting to receiving a loteprednol drop following the intravitreal injection for the research study. Loteprednol is used as a part of regular medical care at the Vistar Eye Center following intravitreal injections but quantifying the magnitude of pain reduction has not been done yet. Additionally, as of now there is no definitive pain management technique following intravitreal injections. This clinical trial is studying the role of loteprednol (corticosteroid) in reducing pain following intravitreal injections for patients with age-related macular degeneration. Participants will be treated with either loteprednol, or artificial tears following one visit for an intravitreal injection at the Vistar Eye Center to test how effective loteprednol is in pain reduction. Pain levels will be assessed by asking participants over the phone about their pain from a scale of 0 to 10 at 2-hours, 1-day, and 1-week following the intravitreal injection. Intravitreal injections will be performed by the retina surgeon, and phone calls will be done with the research coordinator. Artificial tear and medication usage will also be tracked over a 1-week period.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have age-related macular degeneration and be undergoing intravitreal injections for treatment as defined by a retina specialist.

Exclusion Criteria:

* Dementia
* Report baseline eye pain
* Use topical NSAIDs or steroids
* Patient under 18 years old
* History of corticosteroid responsive elevation in intraocular pressure
* Allergy to Loteprednol or Nepafenac
* Pre-existing chronic pain disorders
* Advanced Glaucoma
* Herpes zoster
* Allergy to local anesthetic or penicillin
* Patients unable to consent on own behalf
* Patients unable to communicate pain
* Pregnancy
* Incarceration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2022-12-22 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Post-Intravitreal Injection Pain | 2-hour Post-Intravitreal Injection
  11-point Numerical Rating Scale (0-10, 0 being the lowest level of pain and 10 being highest level of pain)
Post-Intravitreal Injection Pain | 1-day Post-Intravitreal Injection
  11-point Numerical Rating Scale (0-10, 0 being the lowest level of pain and 10 being highest level of pain)
Post-Intravitreal Injection Pain | 1-week Post-Intravitreal Injection
  11-point Numerical Rating Scale (0-10, 0 being the lowest level of pain and 10 being highest level of pain)

SECONDARY OUTCOMES:
Analgesic Medication Use | 2-hour Post-Intravitreal Injection
  Pill count
Analgesic Medication Use | 1-day Post-Intravitreal Injection
  Pill count
Analgesic Medication Use | 1-week Post-Intravitreal Injection
  Pill count
Artificial Tear Use | 2-hour Post-Intravitreal Injection
  Artificial Tear Drop Count
Artificial Tear Use | 1-day Post-Intravitreal Injection
  Artificial Tear Drop Count
Artificial Tear Use | 1-week Post-Intravitreal Injection
  Artificial Tear Drop Count

CONTACTS AND LOCATIONS:
Overall Officials: Vishak John, MD, Principal Investigator — Vistar Eye Center; Romulo Albuquerque, M.D., Ph.D., Principal Investigator — Vistar Eye Center
Locations (1):
- Vistar Eye Center, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ambati J, Fowler BJ. Mechanisms of age-related macular degeneration. Neuron. 2012 Jul 12;75(1):26-39. doi: 10.1016/j.neuron.2012.06.018. PMID 22794258
- [Background] Amon M, Busin M. Loteprednol etabonate ophthalmic suspension 0.5 %: efficacy and safety for postoperative anti-inflammatory use. Int Ophthalmol. 2012 Oct;32(5):507-17. doi: 10.1007/s10792-012-9589-2. Epub 2012 Jun 16. PMID 22707339
- [Background] Chou R, McDonagh MS, Nakamoto E, Griffin J. Analgesics for Osteoarthritis: An Update of the 2006 Comparative Effectiveness Review [Internet]. Rockville (MD): Agency for Healthcare Research and Quality (US); 2011 Oct. Report No.: 11(12)-EHC076-EF. Available from http://www.ncbi.nlm.nih.gov/books/NBK65646/ PMID 22091473
- [Background] DeCroos FC, Afshari NA. Perioperative antibiotics and anti-inflammatory agents in cataract surgery. Curr Opin Ophthalmol. 2008 Jan;19(1):22-6. doi: 10.1097/ICU.0b013e3282f30577. PMID 18090893
- [Background] El-Harazi SM, Feldman RM. Control of intra-ocular inflammation associated with cataract surgery. Curr Opin Ophthalmol. 2001 Feb;12(1):4-8. doi: 10.1097/00055735-200102000-00002. PMID 11150074
- [Background] Fong R, Cavet ME, DeCory HH, Vittitow JL. Loteprednol etabonate (submicron) ophthalmic gel 0.38% dosed three times daily following cataract surgery: integrated analysis of two Phase III clinical studies. Clin Ophthalmol. 2019 Aug 1;13:1427-1438. doi: 10.2147/OPTH.S210597. eCollection 2019. PMID 31447544
- [Background] Grzybowski A, Told R, Sacu S, Bandello F, Moisseiev E, Loewenstein A, Schmidt-Erfurth U; Euretina Board. 2018 Update on Intravitreal Injections: Euretina Expert Consensus Recommendations. Ophthalmologica. 2018;239(4):181-193. doi: 10.1159/000486145. Epub 2018 Feb 1. PMID 29393226
- [Background] Gundogan FC, Yolcu U, Akay F, Ilhan A, Ozge G, Uzun S. Diabetic Macular Edema. Pak J Med Sci. 2016 Mar-Apr;32(2):505-10. doi: 10.12669/pjms.322.8496. PMID 27182271
- [Background] Kaplan RI, Drinkwater OJ, Lee RH, Chod RB, Barash A, Giovinazzo JV, Gologorsky D, Jansen ME, Rosen RB, Gentile RC. Pain Control after Intravitreal Injection Using Topical Nepafenac 0.3% or Pressure Patching: A Randomized, Placebo-Controlled Trial. Ophthalmol Retina. 2019 Oct;3(10):860-866. doi: 10.1016/j.oret.2019.04.022. Epub 2019 Apr 26. PMID 31221565
- [Background] Kaplan RI, Rosen RB, Gentile RC. Optimizing the Patient Experience and Satisfaction: The Role of Topical NSAIDs with Intravitreal Injections. Ophthalmol Retina. 2020 May;4(5):459-460. doi: 10.1016/j.oret.2020.03.004. No abstract available. PMID 32381252
- [Background] Karia N. Retinal vein occlusion: pathophysiology and treatment options. Clin Ophthalmol. 2010 Jul 30;4:809-16. doi: 10.2147/opth.s7631. PMID 20689798
- [Background] Oztas Z, Akkin C, Afrashi F, Nalcaci S. The short-needle intravitreal injection technique. Int J Ophthalmol. 2016 Jun 18;9(6):929-30. doi: 10.18240/ijo.2016.06.24. eCollection 2016. No abstract available. PMID 27366700
- [Background] Popovic MM, Muni RH, Nichani P, Kertes PJ. Topical Nonsteroidal Anti-inflammatory Drugs for Pain Resulting from Intravitreal Injections: A Meta-Analysis. Ophthalmol Retina. 2020 May;4(5):461-470. doi: 10.1016/j.oret.2020.01.024. Epub 2020 Feb 13. PMID 32199867
- [Background] Rifkin L, Schaal S. Shortening ocular pain duration following intravitreal injections. Eur J Ophthalmol. 2012 Nov-Dec;22(6):1008-12. doi: 10.5301/ejo.5000147. Epub 2012 Apr 24. PMID 22562296
- [Background] Shin SH, Park SP, Kim YK. Factors Associated with Pain Following Intravitreal Injections. Korean J Ophthalmol. 2018 Jun;32(3):196-203. doi: 10.3341/kjo.2017.0081. Epub 2018 May 15. PMID 29770638
- [Background] Tan HY, Agarwal A, Lee CS, Chhablani J, Gupta V, Khatri M, Nirmal J, Pavesio C, Agrawal R. Management of noninfectious posterior uveitis with intravitreal drug therapy. Clin Ophthalmol. 2016 Oct 13;10:1983-2020. doi: 10.2147/OPTH.S89341. eCollection 2016. PMID 27789936
- [Background] Toslak D, Thapa D, Chen Y, Erol MK, Paul Chan RV, Yao X. Wide-field fundus imaging with trans-palpebral illumination. Proc SPIE Int Soc Opt Eng. 2017 Jan 28;10045:100451X. doi: 10.1117/12.2252491. Epub 2017 Feb 8. PMID 28781409
- [Background] Williamson A, Hoggart B. Pain: a review of three commonly used pain rating scales. J Clin Nurs. 2005 Aug;14(7):798-804. doi: 10.1111/j.1365-2702.2005.01121.x. PMID 16000093
- [Background] Yahalomi T, Hecht I, Lagstein O, Nemet A, Pe'er L, Hadad F, Keren-Yaar A, Kassem R, Burgansky-Eliash Z, Bar A, Achiron A. REDUCTION OF POSTINTRAVITREAL INJECTION PAIN USING ICE: An Open-Label Interventional Randomized Controlled Trial. Retina. 2020 Jul;40(7):1434-1438. doi: 10.1097/IAE.0000000000002608. PMID 31305506
- See also: Lotemax Information — https://www.rxlist.com/lotemax-side-effects-drug-center.htm